CLINICAL TRIAL: NCT00044447
Title: A Double-Blind, Placebo-Controlled, Parallel Group Comparison Study to Evaluate the Role of the Addition of Amaryl to NIDDM Patients Not Responding to Maximum Dose Metformin and Thiazolidinedione Therapy
Brief Title: Evaluate the Role of Adding Amaryl to Non-Insulin Dependent Diabetes Mellitus Patients Unresponsive to Maximum Dose Metformin & Thiazolidinedione
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HOE490/4033
Record Dates: First submitted 2002-08-28; First posted 2002-08-30 (Estimated); Last update posted 2008-06-19 (Estimated); Status verified 2008-06

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride

INTERVENTIONS:
Drug: Glimepiride

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Amaryl when added to Metformin and Thiazolidinedione (TZD) in non-insulin dependent diabetes mellitus (NIDDM) patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have given their signed informed consent.
* Males or females between 18 and 80 years old. Female patients must be surgically sterile, post-menopausal, or using an accepted method of birth control (i.e., oral contraceptives, intrauterine device, Norplant® system, Depo Provera®, or a spermicide and condom). Female patients of childbearing potential must have a negative serum pregnancy test and be advised not to become pregnant during the study.
* At least 1 year history of NIDDM and performing home blood glucose monitoring.
* Patients must have BMI of > 26 to < 42 kg/m2 at baseline (week 0).
* Patients must have HbA1C > 7.5% but < 9.5% at screen (week -4).
* Patients must have evidence of insulin secretory capacity (fasting C-peptide concentration > or equal to 0.27 nmol/l during the stabilization period).
* Patients must have FPG > 130 mg/dl but < 235 mg/dl prior to (within 48-72 hours) randomization at Visit 1 Week 0.
* Patients must be receiving as their current diabetic therapy stable doses of metformin (at dose of 1.0-2.5gm/day), or metformin extended release at a maximum dose of 2 gm/day and a half maximum to a maximum dose of thiazolidinedione for at least 3 months.
* Patients must be able to understand and willing to adhere to and be compliant with the study protocol.

Exclusion Criteria:

* Patients who require insulin therapy or are currently on other sulfonylureas.
* Patients with a history of hypersensitivity to sulfonylureas.
* Patients with past history of severe hypoglycemia reaction on their current antidiabetic therapy requiring medical attention.
* Patients with a history of acute metabolic complications such as hyperosmolar coma or ketonuria.
* Patients with clinically significant abnormal baseline laboratory values (hematology, blood chemistry or urinalysis) which define a disease or condition, which in the opinion of the investigator may either put the patient at risk because of participation in the study, or may influence the results of the study, or the patient's ability to participate and complete the study. Should there be a laboratory value which, upon initial screening, is substantially outside the normal range, the test should be repeated.
* Patients who had an increase in their thiazolidinedione medication within 2 months of entering the study (Visit 0).
* Patients who had an increase in the metformin medication within 1 month of entering the study (Visit 0).
* Patients whose body weight has changed more than 2% for patients < 250 pounds or 3% for patients >= 250 pounds, during the 4 week stabilization period when compared to the weight at the screening visit 0 (week - 4).
* Patients with acute infections.
* Patients who have received any drug (i.e. a chemotherapy agent) with a well-defined potential for toxicity to a major organ system during the three months prior to the study.
* Patients with clinically significant renal or hepatic disease (i.e. ALT > 2.5 x upper limit of normal) or gastrointestinal disorders that may interfere with absorption of the study drugs.
* Patients who are allergic to sulfonamides and excipients.
* Patients with any history of alcohol or drug abuse.
* Pregnant or lactating females will be excluded.
* Patients with a history of psychosis, emotional or intellectual problems that could impair the ability of the patient to participate in the study or to complete the study.
* Patients who have participated in any investigational study within 30 days prior to Visit 0.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2001-05; Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Change in HbA1C from baseline to Week 26.

SECONDARY OUTCOMES:
Incidence of hypoglycemia.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Dallas Diabetes & Endocrine Center, Dallas, Texas, United States

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com